CLINICAL TRIAL: NCT07108582
Title: Evaluation of the Impact of a Strategy of Perioperative NSAID Suppression in Patients Undergoing Video-assisted Thoracic Surgery (VATS) on the Presence of Chronic Postoperative Pain (CPOP): a Randomised Clinical Trial
Brief Title: Reducing Chronic Pain After Lung Surgery: A Trial of Limiting NSAIDs During Recovery
Acronym: EVADRAINS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9797
Record Dates: First submitted 2025-06-24; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Chronic Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: phase 3, double-blind, multicentre, placebo-controlled, randomised, parallel-arm trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AINS+ (Active Comparator): * 100 mg ketoprofen LP orally administered 30 minutes before surgery,
  * 50 mg ketoprofen intravenously at the end of surgery
  * then 100 mg ketoprofen LP PO twice a day for 7 days following surgery
  Interventions: Drug: protocol for administering NSAIDs already used in routine care
- AINS- (Experimental): no NSAID but a placebo with identical galenic formulations to maintain blindness at all times during participation in the study
  Interventions: Drug: no NSAID

INTERVENTIONS:
Drug: no NSAID — no NSAID but a placebo with identical galenic formulations to maintain blindness at all times during participation in the study
  Arms: AINS-
Drug: protocol for administering NSAIDs already used in routine care — * 100 mg ketoprofen LP orally administered 30 minutes before surgery,
  * 50 mg ketoprofen intravenously at the end of surgery
  * then 100 mg ketoprofen LP PO twice a day for 7 days following surgery
  Arms: AINS+

SUMMARY:
Chronic postoperative pain (CPOP) after video-assisted thoracic surgery (VATS) is severe because it results from lesions at multiple levels: incisions, pulmonary or nerve contusions. PCOD is defined by the IASP (International Association for the Study of Pain) as persistent pain 3 months after surgery. It affects around 30% of patients and significantly impairs recovery and quality of life.

One of the many factors contributing to the appearance of PCOD is acute perioperative pain. To combat this acute pain and limit postoperative chronic pain, a multimodal analgesia strategy is necessary, particularly during thoracic surgery with a high nociceptive potential. This type of protocol will enable acute pain to be controlled by various means: tier 1 analgesics (paracetamol, NSAIDs), tier 2 (nefopam, tramadol) and tier 3 (opioid drugs), locoregional anaesthesia, co-analgesics and non-medicinal techniques. Thus, avoiding NSAIDs will have no effect on the increase in acute pain. A study of the impact of eliminating NSAIDs on chronic pain can therefore be carried out without increasing patients' acute pain.

A team from McGill University, Montreal, Canada, recently discovered a paradoxical effect of anti-inflammatory drugs on the chronicisation of pain. They demonstrated that although anti-inflammatory drugs initially had an acute analgesic effect, they induced neutrophil depletion and a drastic change in the transcriptome postoperatively, leading to more chronic pain. These studies highlight the fact that although NSAIDs have an acute analgesic effect, their use could ultimately prove counterproductive by encouraging the development of CD. However, to date there are no studies demonstrating that a minimum dose or duration of NSAID treatment leads to the development of DCPO. On the basis of these results, it is justified to assess the impact of NSAIDs widely used in routine care in thoracic surgery on the development of DCPO.

In order to improve pain management in the intraoperative phase, nociception monitoring is necessary. The PMD200® (Medasense Biometrics Ltd.) is the most recent monitor designed for this purpose, having demonstrated sensitivity and specificity in detecting nociceptive stimuli under general anaesthesia (4). It will make it possible to guide the administration of analgesic agents by displaying a nociception index (NOL index).

Our hypothesis, based on this work, is that anti-inflammatory drugs, despite having an acute analgesic effect, could promote the development of DCPO after VATS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 to 75
* Patients scheduled for video-assisted thoracic surgery
* Able to give informed consent to participate in the study
* Affiliated to a social health insurance scheme

Exclusion Criteria:

* History of renal insufficiency or chronic pain
* Surgical contraindications to NSAIDs (talc surgery)
* Contraindications to NSAIDs described in the VIDAL RCP (renal insufficiency, allergy, etc.)
* History of chronic use of opioids or anti-inflammatories (continuous use for more than 3 months in the year preceding surgery)
* Urgent surgery;
* Participation in another interventional drug clinical trial.
* Impossibility of giving the subject informed information in the event of difficulties in understanding the subject
* Incapacitated subject (subject to a legal protection measure: safeguard of justice, curatorship, guardianship, future protection mandate, family habilitation)
* Pregnant or breast-feeding

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Postoperative Pain at 3 Months Using a Numerical Rating Scale (NRS) | 3 months post-op

SECONDARY OUTCOMES:
Assessment of Maximum Pain Scores at Rest and During Mobilisation Using a Numerical Rating Scale | Days 0, 1, 3, 1 month and 3 months post-op
Assessment of Neuropathic Pain Using the DN4 Questionnaire | Days 1, 3, 1 month and 3 months post-op
Cumulative Morphine Equivalent Dose of Opioids Administered Intraoperatively | Days 1, 3, 1 month and 3 months post-op
Length of Hospital Stay in Both Patient Groups | up to 3 months post-op
QoR-15 Score | 1 month and 3 months post-op
Collection of Adverse Events and Serious Adverse Events | up to 3 months post-op
Global Proteomic and Transcriptomic (RNA-seq) Analysis and Targeted RT-qPCR of Blood Samples | Days 1, 3 and 3 months post-op
Blood tests for Complete Blood Count by cytometry | Days 0, 1, and 3 months post-op
  Erythrocytes, leukocytes, thrombocytes and associated indices (haemoglobin, haematocrit, etc.)
SF-36 Score | 1 month and 3 months post-op
Physical and Mental Component Scores | 1 month and 3 months post-op
Inflammatory Marker Assessment Including Interleukins | Days 0, 1, and 3 months post-op
Blood tests for C-reactive protein by immunoassay | Days 0, 1, and 3 months post-op
  The results are expressed in mg/L (milligrams per litre)

IPD SHARING:
Plan to Share IPD: Undecided